CLINICAL TRIAL: NCT02372903
Title: Pilot Study About Efficacy of Palmitoylethanolamide-polydatin Combination on Chronic Pelvic Pain in Patients With Laparoscopic Diagnosis of Endometriosis
Brief Title: Efficacy of Palmitoylethanolamide-polydatin Combination on Chronic Pelvic Pain in Patients With Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PELV_25
Record Dates: First submitted 2015-02-13; First posted 2015-02-26 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Endometriosis; Chronic Pelvic Pain
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endometriosis (Experimental): Symptomatic patients with laparoscopic diagnosis of endometriosis
  Interventions: Drug: Administration of micronized Palmitoylethanolamide (PEA)- Transpolydatin

INTERVENTIONS:
Drug: Administration of micronized Palmitoylethanolamide (PEA)- Transpolydatin — Palmitoylethanolamide 600 mg twice daily for 10 days sublingually and oral palmitoylethanolamide 400 mg and polydatin 40 mg, twice daily for 90 days

SUMMARY:
One of the main symptoms of endometriosis is pain, but his pathogenesis is not fully understood. The detection of mast cells in the endometriosis lesions supports the hypothesis that mast cell degranulation may contribute to development of pain and hyperalgesia.

N-acylethanolamines (NAEs) are a class of endogenous compounds that regulate inflammation and pain, controlling mast-cell activation. The aim of the study is to investigate the efficacy of palmitoylethanolamide-polydatin combination on pain relief in symptomatic patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50 years;
* pain visual analog scale (VAS) score>4
* laparoscopic diagnosis of endometriosis (performed in the last three years),
* no assumption of any drugs (in particularly estro-progestinic, progestinic, gonadotropin-releasing hormone (GnRH) agonists and antagonists)
* persistence of symptoms by at least one month

Exclusion Criteria:

* presence of other associated diseases
* assumption of drugs
* menopause
* pregnancy
* unable or unwilling to give written consent patients
* adverse reaction or hypersensitivity to active substance or excipients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change of Pelvic pain as measured by visual analogue scale | Change from Baseline Pelvic Pain at 90 days of treatment

SECONDARY OUTCOMES:
Change of Pelvic pain as measured by visual analogue scale | Change from baseline Pelvic Pain after 30 days from the suspension of the therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department,, Monserrato, Cagliari, Italy